CLINICAL TRIAL: NCT04354259
Title: Interferon Lambda for Immediate Antiviral Therapy at Diagnosis (ILIAD): A Phase II Randomized, Double-blind, Placebo-controlled, Multicenter Trial to Evaluate the Effect of Peginterferon Lambda for the Treatment of COVID-19
Brief Title: Interferon Lambda for Immediate Antiviral Therapy at Diagnosis in COVID-19
Acronym: ILIAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Michael Garron Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-5334
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Sars-CoV2; Covid-19
Keywords: peginterferon lambda
MeSH Terms: conditions — COVID-19 | interventions — peginterferon lambda-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Ambulatory Cohort - Treatment (Experimental): to receive a single dose of peginterferon lambda 180µg SC at baseline (day 0).
  Interventions: Drug: Peginterferon Lambda-1A
- Ambulatory Cohort - placebo (Placebo Comparator): Patients in the arm will be given a single injection of 0.9% sodium chloride (normal saline) solution at baseline (day 0). A plastic 1 mL syringe will be prefilled by the study pharmacy. Each syringe will contain 0.5 mL (0.45 mL to match the volume of the Interferon plus 0.05 mL overfill) to allow for needle priming by the unblinded study nurse.
  Interventions: Other: placebo
- Hospitalized Cohort - Treatment (Experimental): To receive a dose of peginterferon lambda 180µg SC at baseline and a second dose on day 5.
  Interventions: Drug: Peginterferon Lambda-1A
- Hospitalized Cohort - placebo (Placebo Comparator): Patients in the arm will be given an injection of 0.9% sodium chloride (normal saline) solution at baseline (day 0). A plastic 1 mL syringe will be prefilled by the study pharmacy. Each syringe will contain 0.5 mL (0.45 mL to match the volume of the Interferon plus 0.05 mL overfill) to allow for needle priming by the unblinded study nurse. Patients will be administered a second dose of placebo on day 5.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Peginterferon Lambda-1A — Peginterferon lambda is a covalent conjugate of human recombinant non-pegylated IFN lambda (IFN L) and a 20-kDa linear PEG chain. Peginterferon lambda Injection is a sterile, nonpyrogenic, ready-to-use solution (0.4 mg/mL) that is clear to opalescent, colorless to pale yellow, and essentially free of particles. Lambda Injection is provided in a 1-mL long Type I glass syringe (0.18 mg/syringe) with a staked 29-gauge, 1/2- inch, thin-walled needle. The syringe has a rigid needle shield and is stoppered with a plunger stopper. Syringes are prefilled with a solution of Peginterferon lambda Injection, mannitol, L-histidine, polysorbate 80, hydrochloric acid, and water for injection; they are intended for a single use at adjustable doses. The syringe is marked with dose indicator lines, which are used as a reference point for administering the correct dose.
  Arms: Ambulatory Cohort - Treatment; Hospitalized Cohort - Treatment
Other: placebo — injection of 0.9% sodium chloride (normal saline) solution. A plastic 1 mL syringe will be prefilled by the study pharmacy. Each syringe will contain 0.5 mL (0.45 mL to match the volume of the Interferon plus 0.05 mL overfill) to allow for needle priming by the unblinded study nurse.
  Arms: Ambulatory Cohort - placebo; Hospitalized Cohort - placebo

SUMMARY:
Interferon lambda is one of the main arms of the innate antiviral immune response and is critical for controlling respiratory viral infections in mice. Interferon lambda has a better side effect profile than other interferons because of the limited tissue distribution of its receptor. Peginterferon lambda is a long-acting form that has been studied extensively in human trials in viral hepatitis, confirming its safety. We propose to evaluate peginterferon-lambda in ambulatory and hospitalized patients with mild to moderate COVID-19.

DETAILED DESCRIPTION:
The study uses an adaptive design with initial enrolment in the Ambulatory cohort (Cohort A) followed by a safety assessment before initiation of enrolment in the Hospitalized cohort (Cohort B).

Ambulatory patients (Cohort A) with confirmed COVID-19 deemed well enough for home isolation will be randomized to receive a single subcutaneous injection of Peginterferon lambda 180µg or saline placebo prior to discharge. Patients will be followed remotely with visits for a repeat swab at Day 3 and 7 with the primary endpoint being the proportion positive for SARS-CoV-2 on Day 7.

Safety data will be reviewed by the Data Safety and Monitoring Committee after 50% of the Ambulatory cohort (n=60) has been enrolled. If the committee approves study continuation, enrolment will continue in the Ambulatory cohort (Cohort A) and will begin in the Hospitalized cohort (Cohort B).

Hospitalized patients (Cohort B) with moderate but not severe COVID-19 will be enrolled and randomized to Peginterferon lambda 180µg or saline placebo on Day 0 and 5. The primary endpoint will be clinical outcomes on the WHO ordinal scale. In addition to the primary endpoint on which the study is powered, numerous secondary endpoints will be evaluated. Samples will also be collected for ancillary studies to better understand predictors of disease severity and response to treatment.

ELIGIBILITY:
Cohort A - Ambulatory

Inclusion Criteria

1. Adult patients between the ages of 18 and 75 years.
2. Confirmed COVID-19 infection by PCR within 7 days of symptom onset (fever, respiratory symptoms, sore throat).
3. Discharged to home isolation.
4. Willing and able to sign informed consent.
5. Willing and able to follow-up by daily phone or videoconference.
6. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal. Adequate methods of contraception are:

   a. For female patients i. Hormonal contraceptives including progestogen injection (eg, Depo-Provera®), combined oral contraceptive pill or vaginal ring for ≥ 3 months before screening AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or ii. Intrauterine device (IUD) or intrauterine system (IUS) in place ≥ 3 months before screening AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or iii. Surgical sterilization of the partner (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or iv. Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening.

   b. For male patients i. Surgical sterilization (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom or diaphragm with spermicide or cervical cap with spermicide) from screening, or ii. Consistently and correctly use a condom from screening AND female partner must agree to use a hormonal contraceptive, a nonhormonal nonbarrier method (eg, copper IUD), or a nonhormonal barrier method (eg, diaphragm with spermicide or cervical cap with spermicide).

Exclusion Criteria

1. Requirement for hospital admission
2. Current immunosuppression due to medication (steroids, biologics, chemotherapy) or underlying condition such as organ/bone marrow transplant or untreated HIV or HIV infection with detectable HIV RNA and/or CD4 count of <500.
3. Pregnancy (or positive urine pregnancy test) or lactating
4. The following pre-existing medical conditions:

   1. Known seizure disorder
   2. Known retinal disease requiring therapy
   3. Known autoimmune condition requiring therapy more intensive than intermittent non-steroidal anti-inflammatories in the prior 6 months (rheumatoid arthritis, lupus, inflammatory bowel disease)
   4. Known history of chronic obstructive pulmonary disease (COPD) or asthma associated with functional impairment
   5. Known cirrhosis with any history of decompensation (ascites, variceal bleeding or hepatic encephalopathy)
   6. Known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis
   7. Severe psychiatric disorder - schizophrenia, bipolar disorder, depression with prior suicidality
   8. Any other underlying medical (cardiac, liver, renal, neurological, respiratory) or psychiatric condition that in the view of the investigator would preclude use of peginterferon lambda
5. Advanced cancer or other illness with life expectancy of < 1 year
6. Known alcohol or drug dependence that in the opinion of the investigator would impair study participation
7. Known prior intolerance to interferon treatment
8. Enrolment in another clinical trial with use of any investigational agent in the prior 30 days
9. Use of off-label therapy for COVID-19

Cohort B - Hospitalized

Inclusion Criteria

1. Adult patients over age 18
2. SARS-CoV-2 RNA-positive on nasopharyngeal swab/respiratory specimen within 10 days of symptom onset
3. Admitted to hospital for management of COVID-19
4. Willing and able to provide informed consent
5. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal. Adequate methods of contraception are:

   a. For female patients: i. Hormonal contraceptives including progestogen injection (eg, Depo-Provera®), combined oral contraceptive pill or vaginal ring for ≥ 3 months before screening AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or ii. Intrauterine device (IUD) or intrauterine system (IUS) in place ≥ 3 months before screening AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or iii. Surgical sterilization of the partner (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or iv. Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening.

   b. For male patients: i. Surgical sterilization (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom or diaphragm with spermicide or cervical cap with spermicide) from screening, or ii. Consistently and correctly use a condom from screening AND female partner must agree to use a hormonal contraceptive, a nonhormonal nonbarrier method (eg, copper IUD), or a nonhormonal barrier method (eg, diaphragm with spermicide or cervical cap with spermicide).

Exclusion Criteria

1. Severity of illness

   1. Respiratory failure (requiring>6L O2 or intubation in the ER)
   2. Shock - systolic BP<90 mmHg or mean arterial BP<60 mmHg after fluid resuscitation
2. Pregnancy (or positive urine pregnancy test) or lactating
3. The following pre-existing medical conditions:

   1. Known seizure disorder
   2. Known retinal disease requiring therapy
   3. Known autoimmune condition requiring therapy more intensive than intermittent non-steroidal anti-inflammatories in the prior 6 months (rheumatoid arthritis, lupus, inflammatory bowel disease)
   4. Known cirrhosis with any history of decompensation (ascites, variceal bleeding or hepatic encephalopathy)
   5. Known chronic kidney disease with estimated creatinine clearance < 30 mL/minute or need for dialysis
   6. Severe psychiatric disorder - uncontrolled schizophrenia, bipolar disorder, depression with prior suicidality
   7. Any other underlying medical (cardiac, liver, renal, neurological, respiratory) or psychiatric condition that in the view of the investigator would preclude use of peginterferon lambda
4. Known prior intolerance to interferon treatment
5. Enrolment in another clinical trial with use of an antiviral agent in the prior 30 days (co-enrollment with immunomodulatory agents permitted)
6. Use of off-label therapy for COVID-19
7. Any of the following abnormal laboratory indices

   1. Hemoglobin < 100 mg/dL
   2. Platelet count < 75,000 cells/mm3
   3. Absolute neutrophil count < 1,000 cells/mm3
   4. Estimated creatinine clearance < 30 cc/mL
   5. Total bilirubin > 2x upper limit of normal (ULN)
   6. Alanine aminotransferase (ALT) > 5x ULN
   7. Aspartate aminotransferase (AST) > 5x ULN
   8. Lipase or amylase > 2x ULN
   9. Random blood glucose > 20 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Cohort A (Ambulatory) - Proportion swab negative at day 7 (Primary efficacy endpoint) | At day 7
  The proportion of participants with negative SARS-CoV-2 RNA on nasopharyngeal swab.
Cohort A (Ambulatory) - Treatment-emergent and treatment related serious adverse events (Primary Safety Endpoint) | Day 0 to Day 28
  The rate of treatment-emergent and treatment-related serious adverse events (SAEs)
Cohort B (Hospitalized) - Ordinal Scale (Primary Efficacy Endpoint) | At Day 14
  Clinical status on an ordinal scale at Day 14
Cohort B (Hospitalized) - treatment-emergent and treatment-related serious adverse events (Primary Safety Endpoint) | Day 0 to Day 28
  The rate of treatment-emergent and treatment-related serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cohort A (Ambulatory) - Symptom Resolution (Clinical Outcome #1) | Day 0 to Day 14
  Time to resolution of symptoms (fever, cough, diarrhea)
Cohort A (Ambulatory) - Symptom severity scores (Clinical Outcome #2) | Day 0 to Day 7
  Change in relative categorical symptom scores (respiratory, gastrointestinal, fever) - none, mild, moderate, severe and no change, worse, better
Cohort A (Ambulatory) - Hospitalization (Clinical Outcome #3) | Day 0 to Day 14
  Proportion with need for hospital admission
Cohort A (Ambulatory) - Adverse and serious adverse events (Clinical Outcome #4) | Day 0 to Day 14
  Adverse events and serious adverse events
Cohort A (Ambulatory) - Swab negative at day 3 (Virologic/Immunological Outcome #1) | At Day 3
  Proportion negative for SARS-CoV-2 RNA by nasopharyngeal swab
Cohort A (Ambulatory) - Time RNA negativity (Virologic/Immunological Outcome #2) | Day 0 to Day 14
  Time to SARS-CoV-2 RNA negativity on mid-turbinate nasal swab or saliva
Cohort A (Ambulatory) - Proportion viremic (Virologic/Immunological Outcome #3) | Day 0 and Day 7
  Proportion with SARS-CoV-2 RNA in blood.
Cohort A (Ambulatory) - Proportion with antibodies (Virologic/Immunological Outcome #4) | Day 0 and Day 7
  Proportion with SARS-CoV-2 antibodies blood
Cohort A (Ambulatory) - Correlation with interferon lambda 4 genotype (Virologic/Immunological Outcome #5) | Through day 7
  Correlation of virologic response with interferon lambda 4 (IFNL4) genotype
Cohort A (Ambulatory) - Symptoms in household contacts (Transmission Outcome #1) | Day 0 to Day 14
  Proportion with symptom development in household contacts (categorical symptom type yes/no)
Cohort A (Ambulatory) - COVID-19 in household contacts (Transmission Outcome #2) | At Day 30
  Proportion with confirmed diagnosis of COVID-19 in household contacts
Cohort B (Hospitalized) - Ordinal scale (Clinical Outcome #1) | At Days 7, 21 and 28
  Clinical status on the ordinal scale
Cohort B (Hospitalized) - ICU admission (Clinical Outcome #2) | Day 0 to day 28
  Proportion with ICU admission during hospitalization
Cohort B (Hospitalized) - Need for intubation (Clinical Outcome #3) | Day 0 to Day 14 and to Day 28
  Proportion with need for intubation
Cohort B (Hospitalized) - Length of hospital stay (Clinical Outcome #4) | Day 0 to Day 14
  Length of hospital stay (days)
Cohort B (Hospitalized) - Change in respiratory symptom score (Clinical Outcome #5) | Day 0 to 7, Day 0 to 14, and Day 0 to 28
  Change in respiratory symptom score (score 0 to 7 with higher scores indicating more severe disease)
Cohort B (Hospitalized) - All-cause mortality (Clinical Outcome #6) | At day 28 and day 90
  All-cause mortality
Cohort B (Hospitalized) - Readmission to hospital (Clinical Outcome #7) | From Day 0 -28 and from Day 0 - 90
  Proportion with readmission to hospital
Cohort B (Hospitalized) - COVID-19-related mortality (Clinical Outcome #8) | At day 28
  COVID-19-related mortality
Cohort B (Hospitalized) - Adverse (AEs) and Serious Adverse Events (SAEs) (Clinical Outcome #9) | Day 0 to day 28
  Adverse (AEs) and Serious Adverse Events (SAEs)
Cohort B (Hospitalized) - Dose reduction or dose omission (Clinical Outcome #10) | Day 5 to day 9
  Frequency of dose reduction or dose omission for the second dose of peginterferon lambda
Cohort B (Hospitalized) - Time to viral negativity (Virologic/Immunological Outcome #1) | Day 0 - Day 28
  Time to SARS-CoV-2 RNA negativity.
Cohort B (Hospitalized) - Proportion negative swab. (Virologic/Immunological Outcome #2) | Days 0-7, 10, 12, 14, 18, 21, 25 and 28
  Proportion negative for SARS-CoV-2 RNA by mid-turbinate swab
Cohort B (Hospitalized) - Quantitative viral load by nasal swab (Virologic/Immunological Outcome #3) | Day 0 - Day 28
  Change in quantitative SARS-CoV-2 RNA by mid-turbinate swab over time
Cohort B (Hospitalized) - Correlation with interferon lambda 4 (IFNL4) genotype (Virologic/Immunological Outcome #4) | Through Day 14
  Correlation of virologic response with interferon lambda 4 (IFNL4) genotype
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #5) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in hemoglobin over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #6) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in white blood cell count over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #7) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in lymphocyte count over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #8) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in platelet count over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #9) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in ALT over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #10) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in AST over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #11) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in ALP over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #12) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in bilirubin over time.
Cohort B (Hospitalized) - Safety Markers (Virologic/Immunological Outcome #13) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in albumin over time.
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #14) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in ferritin over time.
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #15) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in lactate dehydrogenase over time.
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #16) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in c-reactive protein over time
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #17) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in D-dimers over time.
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #18) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in creatine kinase over time.
Cohort B (Hospitalized) - Inflammatory Markers (Virologic/Immunological Outcome #19) | From Day 0 - Day 7 and to Day 14, 21, and 28
  Change in troponin over time.
Cohort B (Hospitalized) - Proportion with Antibody (Virologic/Immunological) Outcome #20) | At Day 7, 14, 21, and 28
  Proportion with SARS-CoV-2 Antibody.
Cohort B (Hospitalized) - Proportion with viremia (Virologic/Immunological Outcome #21) | Day 0, Day 7, 14, 21, and 28
  Proportion with SARS-CoV-2 RNA in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Feld, MD, Principal Investigator — University Health Network, Toronto
Locations (7):
- Brazil (3):
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital das Clínicas São Paulo, São Paulo
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feld JJ, Kandel C, Biondi MJ, Kozak RA, Zahoor MA, Lemieux C, Borgia SM, Boggild AK, Powis J, McCready J, Tan DHS, Chan T, Coburn B, Kumar D, Humar A, Chan A, O'Neil B, Noureldin S, Booth J, Hong R, Smookler D, Aleyadeh W, Patel A, Barber B, Casey J, Hiebert R, Mistry H, Choong I, Hislop C, Santer DM, Lorne Tyrrell D, Glenn JS, Gehring AJ, Janssen HLA, Hansen BE. Peginterferon lambda for the treatment of outpatients with COVID-19: a phase 2, placebo-controlled randomised trial. Lancet Respir Med. 2021 May;9(5):498-510. doi: 10.1016/S2213-2600(20)30566-X. Epub 2021 Feb 5. PMID 33556319
- [Derived] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708
- [Derived] Moschen AR. IBD in the time of corona - vigilance for immune-mediated diseases. Nat Rev Gastroenterol Hepatol. 2020 Sep;17(9):529-530. doi: 10.1038/s41575-020-0333-5. PMID 32555385

DOCUMENTS (1):
  • Study Protocol (2021-01-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT04354259/Prot_000.pdf